CLINICAL TRIAL: NCT01799252
Title: Side Effects and Adherence Associated With Doxycycline Use Following Medical Abortion
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Other Study IDs: 7000
Record Dates: First submitted 2012-12-07; First posted 2013-02-26 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Abortion
Keywords: medical abortion; doxycycline; antibiotics; adherence; nausea
MeSH Terms: conditions — Nausea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Doxy: Women who are prescribed a seven-day regimen of doxycycline following medical abortion
- No Doxy: Women who are not prescribed antibiotics following medical abortion

SUMMARY:
The effectiveness of antibiotic treatment at reducing post-abortion infection is unclear. The experiences of women prescribed routine antibiotics after medical abortion is missing from the existing evidence. This study seeks to add to the literature evidence of the side effects associated with antibiotic treatment that women experience and their adherence to prescribed regimens.

DETAILED DESCRIPTION:
Medical abortion (MA) consists of administering medication, typically a combination of mifepristone and misoprostol, to induce an abortion without any invasive procedures. Early first trimester MA is effective1, highly acceptable to women, and safe. The risk of infection following medical abortion is small, at less than 1%. In rare circumstances, pelvic infection with clostridia bacteria following medical abortion has resulted in death. Since 2000, when mifepristone was registered in the United States, 8 such deaths have been recorded in the US.

Following the publication of case reports of four clostridium-associated deaths after medical abortion in 2005, the reproductive health community reacted swiftly. Medical abortion protocols were altered in an effort to curb these drastic and rapidly fatal infections. Antibiotic treatment, typically a seven-day course of doxycycline, has become widespread in the United States.

The effectiveness of antibiotic treatment at reducing post-abortion infection is unclear. The experiences of women prescribed routine antibiotics after medical abortion is missing from the existing evidence. This study seeks to add to the literature evidence of the side effects associated with antibiotic treatment that women experience and their adherence to prescribed regimens.

ELIGIBILITY:
Inclusion Criteria:

* Women who are having MA at the study clinic and are willing to complete a self-administered, computer-based questionnaire 7-14 days after taking mifepristone
* Women who can read English or Spanish
* In the doxycycline arm: Women who have been prescribed doxycycline

Exclusion Criteria:

* Women who were treated with antibiotics for a medical condition unrelated to their medical abortion between the initial visit and follow-up appointment
* Women who have previously enrolled in this study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll 610 women. Women will be recruited from 5 clinics and will self-administer, or if necessary, a study coordinator will administer, a computer-based questionnaire 7-14 days following administration of mifepristone.
Sampling Method: Non-Probability Sample
Enrollment: 582 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Incidence rates of nausea | 7-14 days following medical abortion
  Compare the incidence rates of nausea between women who are prescribed a seven-day regimen of doxycycline to women who are not prescribed antibiotics following medical abortion
adherence | 7-14 days following medical abortion
  Document the self-reported adherence to antibiotic regimens following medical abortion

SECONDARY OUTCOMES:
Nausea rates | 7-14 days following medical abortion
  Compare the rates of nausea between women who take at least one doxycycline pill to women who do not take any doxycycline following medical abortion
Non-nausea side effects | 7-14 days following medical abortion
  Compare the rates of other (non-nausea) side effects between women who are prescribed a seven-day regimen of doxycycline to women who are not prescribed antibiotics following medical abortion
Additional medications | 7-14 days following medical abortion
  Compare the use of additional medication to treat side effects between women who take antibiotics and women who do not take antibiotics following medical abortion
Cost | at time of filling prescription
  Document the cost to women of antibiotics regimens following medical abortion

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (7):
- United States (7):
  - Feminist Women's Health Center, Atlanta, Georgia
  - Family Planning Associates, Chicago, Illinois
  - Planned Parenthood Mid and South Michigan, Ann Arbor, Michigan
  - Planned Parenthood MN, ND, SD, Saint Paul, Minnesota
  - Family Practice and Sidney Hillman Family Practice at the Institute for Family Health, New York, New York
  - NYU/Bellevue Hospital Center, Women's Health Center, New York, New York
  - Cedar River Clinic, Renton, Washington

REFERENCES:
- [Derived] Frye LJ, Chong E, Winikoff B; NCT01799252 Trial Investigators. What happens when we routinely give doxycycline to medical abortion patients? Contraception. 2015 Jan;91(1):19-24. doi: 10.1016/j.contraception.2014.09.001. Epub 2014 Sep 15. PMID 25444253
- See also: Sponsor website — http://www.gynuity.org